CLINICAL TRIAL: NCT01930604
Title: Botulinum Toxin Treatment in Craniofacial, Inguinal, Palmar, Plantar and Truncal Hyperhidrosis, a Randomized, Double Blind, Placebo Controlled Study
Brief Title: Botulinum Toxin Treatment in Craniofacial, Inguinal, Palmar, Plantar and Truncal Hyperhidrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carl Swartling (Other)
Responsible Party: Sponsor-Investigator, Carl Swartling, MD, PhD, Hidrosis Clinic, Stockholm, Sweden
Organization: Hidrosis Clinic, Stockholm, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTXHH11
Record Dates: First submitted 2013-08-16; First posted 2013-08-29 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Hyperhidrosis
Keywords: Palmar hyperhidrosis.; Plantar hyperhidrosis.; Inguinal (groins and buttocks) hyperhidrosis.; Craniofacial hyperhidrosis.; Truncal hyperhidrosis.
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A; rimabotulinumtoxinB

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Palmar hyperhidrosis, Botox (onabotulinumtoxinA) (Active Comparator): Solution for injection, individual dosing, maximum dose 400 units, single treatment session.
  Interventions: Drug: Botox (onabotulinumtoxinA)
- Palmar hyperhidrosis, NaCl (Placebo Comparator): Solution for injection, individual dosing, injection volume corresponding to active comparator, single treatment session.
  Interventions: Drug: NaCl (placebo)
- Plantar hyperhidrosis, Botox (onabotulinumtoxinA) (Active Comparator): Solution for injection, individual dosing, maximum dose 400 units, single treatment session.
  Interventions: Drug: Botox (onabotulinumtoxinA)
- Plantar hyperhidrosis, NaCl (Placebo Comparator): Solution for injection, individual dosing, injection volume corresponding to active comparator, single treatment session.
  Interventions: Drug: NaCl (placebo)
- Inguinal (groins/buttocks) hyperhidrosis, Botox (ona...) (Active Comparator): Solution for injection, individual dosing, maximum dose 400 units, single treatment session.
  Interventions: Drug: Botox (onabotulinumtoxinA)
- Inguinal (groins/buttocks) hyperhidrosis, NaCl (Placebo Comparator): Solution for injection, individual dosing, injection volume corresponding to active comparator, single treatment session.
  Interventions: Drug: NaCl (placebo)
- Craniofacial hyperhidrosis, NeuroBloc/Myobloc (rima...) (Active Comparator): Solution for injection, individual dosing, maximum dose 2500 units, single treatment session.
  Interventions: Drug: NeuroBloc/Myobloc (rimabotulinumtoxinB)
- Craniofacial hyperhidrosis, NaCl (Placebo Comparator): Solution for injection, individual dosing, injection volume corresponding to active comparator, single treatment session.
  Interventions: Drug: NaCl (placebo)
- Truncal hyperhidrosis, NeuroBloc/Myobloc (rimabotulinumtoxinB) (Active Comparator): Solution for injection, individual dosing, maximum dose 5000 units, single treatment session.
  Interventions: Drug: NeuroBloc/Myobloc (rimabotulinumtoxinB)
- Truncal hyperhidrosis, NaCl (Placebo Comparator): Solution for injection, individual dosing, injection volume corresponding to active comparator, single treatment session.
  Interventions: Drug: NaCl (placebo)

INTERVENTIONS:
Drug: Botox (onabotulinumtoxinA)
  Arms: Inguinal (groins/buttocks) hyperhidrosis, Botox (ona...); Palmar hyperhidrosis, Botox (onabotulinumtoxinA); Plantar hyperhidrosis, Botox (onabotulinumtoxinA)
Drug: NeuroBloc/Myobloc (rimabotulinumtoxinB)
  Arms: Craniofacial hyperhidrosis, NeuroBloc/Myobloc (rima...); Truncal hyperhidrosis, NeuroBloc/Myobloc (rimabotulinumtoxinB)
Drug: NaCl (placebo)
  Arms: Craniofacial hyperhidrosis, NaCl; Inguinal (groins/buttocks) hyperhidrosis, NaCl; Palmar hyperhidrosis, NaCl; Plantar hyperhidrosis, NaCl; Truncal hyperhidrosis, NaCl

SUMMARY:
Hyperhidrosis is defined as excessive sweating and affects about 2.8 % of the population.

It has been shown to have a deleterious effect on the quality of life measured using the Dermatology Life Quality Index (DLQI) which is one of the most widely used dermatology-specific quality of life instruments. This is comparable to the effect on quality of life in patients with severe psoriasis of the skin as well as to nodulocystic acne patients before treatment with oral isotretinoin.

The clinical effect of Botulinum Toxin (Btx) A has been established in three randomized controlled trials (RCT) in axillary hyperhidrosis. One RCT has indicated a positive effect in palmar hyperhidrosis. Although there is increasing evidence that Btx A and B have a similar effect on hyperhidrosis of other parts of the body (ie hyperhidrosis of the face, trunk, groin and feet) which is reported in case-reports and open studies there is still a great need for more controlled studies. This is why we will carry out this randomized, double-blind, placebo-controlled study to investigate the clinical effect and safety of Btx A in palmar, plantar and inguinal (groins/buttocks) hyperhidrosis and the clinical effect and safety of Btx B in craniofacial and truncal hyperhidrosis, respectively. Besides using the DLQI instrument we will also study Btx A/B to elucidate the impact of this treatment on quality of life using a generic instrument, the effect on anxiety and depressive symptoms, sweating, and patients´global assessment of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent received from patient
* Informed consent received from patient´s parents (when patient < 18 years)
* Hyperhidrosis of the head, trunk, groins/buttocks, hands or feet
* Age > 16 years
* Patients must be previously untreated with Btx A/B
* If female, patient is post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom*) throughout the study. If male with a female partner of childbearing potential, willing to use an acceptable method of birth control for the study duration of the study, for both female and male, acceptable birth control must be used for at least 3 months after the last dose of study medication.

  * A condom alone is not considered an acceptable method for birth control. Two barrier methods only are not considered an acceptable method of birth control.
* Patients must have DLQI-score ≥ 10 and HDSS-score ≥ 3

Exclusion Criteria:

* Contraindication to Btx
* Use of aminoglycosides, tetracyclines , spectinomycin, lincomycin, polymyxin or muscle relaxants
* Pregnancy or lactation
* Patients unwilling to meet the requirements of the protocol
* Other medical or social reasons for exclusion at the discretion of the Investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2013-09; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
DLQI (Dermatology Life Quality Index) | 3±1 weeks after treatment
  The primary endpoint is scores on DLQI-values at follow-up in the Btx A/B treatment groups when compared to the placebo groups.

SECONDARY OUTCOMES:
AE (Adverse Events) | Up to 12 weeks
  Safety by recording of reported adverse events (AE) by the patient at the clinic visits
Gravimetry | Before treatment and 3±1 weeks after treatment
  The amount of sweat is measured gravimetrically.
HDSS (Hyperhidrosis Disease Severity Scale) | Before treatment and 3±1 weeks after treatment
Health outcome (EQ-5D) | Before treatment and 3±1 weeks after treatment
LSAS-SR (Liebowitz Social Anxiety Scale-Self Report) | Before treatment and 3±1 weeks after treatment
MADRS-S (Montgomery-Asberg Depression Rating Scale-Self report) | Before treatment and 3±1 weeks after treatment
Global Assessment of Therapy | 3±1 weeks after treatment
  The patient will be asked at the follow-up visit (3±1 weeks after treatment) to give his/her subjective opinion and rate the effect of the treatment using a scale ranging from 1-5.
DLQI (Dermatology Life Quality Index) | Before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carl Swartling, MD, PhD, Principal Investigator — Hidrosis Clinic, Warfvinges väg 35, Stockholm, Sweden
Locations (1):
- Carl Swartling, Stockholm, Sweden